CLINICAL TRIAL: NCT00244634
Title: A Dose-Ranging and Safety Study of Candesartan Cilexetil in Hypertensive Pediatric Subjects 6 to <17 Years of Age: A 4-Week, Multinational, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study
Brief Title: Atacand Dose Range Finding Study in Pediatric Subjects 6 to <17 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D2451C00261; 261A
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2007-12-19 (Estimated); Status verified 2007-12

CONDITIONS: Pediatric Hypertension

INTERVENTIONS:
Drug: candsartan cilexetil

SUMMARY:
Study 261A is a dose-ranging and safety study of candesartan cilexetil. It is a multinational, multicenter, randomized, double-blind, placebo-controlled, parallel-group study with a 4 week treatment period in hypertensive pediatric subjects.

Subjects undergo a screening evaluation, then a 1-week, single-blind, placebo run-in after which eligible subjects are allocated to receive 1 of 3 dose levels of candesartan cilexetil or placebo. The study includes 2 panels based on subject weight.

The primary efficacy analysis is based on the intent-to-treat population and tests for slope = 0 in a linear regression model with change in sitting systolic blood pressure as the dependent and non-zero dose pooled across weight panels as the independent variable. For subjects without a Double-Blind Week 4 blood pressure determination, carrying the last value forward assigns the value.

Additional analyses will include data pooled from a similar dose ranging study conducted in children 1 to < 6 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 6 to < 17 years-of-age after parent or guardian's signing of informed consent.

Subjects with hypertension that is either:

* Diagnosed and untreated with a mean sitting systolic and/or diastolic blood pressure ≥ 95th percentile and ≤ 20 mm Hg (systolic) and/or 10 mm Hg (diastolic) above the 95th percentile at randomisation based on height-adjusted charts for age and gender; or
* Previously diagnosed and currently treated with mean sitting systolic blood pressure and/or diastolic blood pressure ≥ 95th percentile and ≤ 20 mm Hg (systolic) and/or 10 mm Hg (diastolic) above the 95th percentile at randomisation (off treatment) based on height-adjusted charts for age and gender.

Females of childbearing potential (post-menarche) must have a negative urine pregnancy test prior to randomization and adhere to a pregnancy prevention method (abstinence, barrier method plus spermicidal foam, oral, or implanted contraceptive).

A signed informed consent by a parent or a legal guardian and an assent form signed by the subject (if applicable).

Exclusion Criteria:

* Any situation, clinical condition or laboratory abnormality that, in the opinion of the investigator or sponsor, may interfere with the subject's participation in the study or would pose a significant risk to the subject or interfere with the assessment of safety and efficacy endpoints.
* Hypertension secondary to coarctation of the aorta, pheochromocytoma, hyperthyroidism, Cushing's syndrome, or medications (eg: corticosteroids).
* Known history of bilateral renal artery stenosis, unilateral renal artery stenosis or a renal transplant.
* Glomerular filtration rate < 50 mL/min based on an estimated value using the Schwartz Formula.
* Nephrotic syndrome not in remission.
* Insulin dependent diabetes mellitus.
* Known bleeding, coagulation, or platelet disorder that could interfere with blood sampling.
* Clinically significant valvular heart disease.
* Clinical diagnosis of heart failure.
* Clinically significant arrhythmia (eg, any arrhythmia requiring medical therapy or that causes symptoms).
* Second or third degree AV block.
* Pregnant or breast-feeding an infant.
* Impaired liver function defined as either acute liver disease or chronic liver disease with persistent liver enzyme values greater than 1½ times the upper limit of the reference range for AST or ALT.
* Known hypersensitivity to ARBs.
* Unable to be off antihypertensive medication (diuretics, beta blockers, ACE Inhibitors, etc) for 6-weeks.
* Inability to discontinue medications which may contribute to elevated blood pressure e.g. systemic corticosteroids.
* Currently using, or used within 14 days prior to receiving double-blind medication, any concomitant medications which in the opinion of the investigator could negatively affect the subject.
* Unable or unwilling to comply with the study requirements including blood sampling and swallowing study drug tablets.
* Received an investigational agent within 30 days prior to receiving study medication.
* Alcohol or drug abuse.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 238
Dates: Start 2003-09; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Trough sitting systolic blood pressure, the measure of effect is change from baseline to double-blind Week 4.
The endpoint (outcome variable) is the slope by linear regression

SECONDARY OUTCOMES:
To further evaluate the antihypertensive effects and the safety of candesartan cilexetil in hypertensive pediatric subjects.
Determine the slope of the change from baseline to double-blind treatment in:
• trough sitting diastolic blood pressure,
• trough standing diastolic blood pressure and standing systolic blood pressure,
• trough sitting pulse pressure.
- Mean change from baseline in SiSBP, SiDBP, pulse pressure, and standing SBP and DBP relative to placebo for each dose group and for all dose groups pooled
- Safety as assessed by adverse events, adverse events that necessitate study drug discontinuation, SAEs, heart rate, electrocardiographic findings, physical exam findings, and laboratory tests.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Atacand Medical Science Director, MD, Study Director — AstraZeneca
Locations (44):
- United States (36):
  - Research Site, Beverly Hills, California
  - Research Site, Los Angeles, California
  - Research Site, Madera, California
  - Research Site, Yuba City, California
  - Research Site, Newark, Delaware
  - Research Site, Wilmington, Delaware
  - Research Site, Miami, Florida
  - Research Site, Athens, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Ann Arbor, Michigan
  - Research Site, Jackson, Mississippi
  - Research Site, Port Gibson, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Paterson, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, New Hyde Park, New York
  - Research Site, The Bronx, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Beaumont, Texas
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Charleston, West Virginia
- Research Site, Ghent, Belgium
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Miskolc
  - Research Site, Szeged
- Slovakia (4):
  - Research Site, Bratislava
  - Research Site, Martin
  - Research Site, Myjava
  - Research Site, Trnava